CLINICAL TRIAL: NCT03271164
Title: Prospective Randomized Controlled Case Series Evaluating the Safety and Efficacy of FBPM10 System When Compared to Standard of Care in the Treatment of Post-surgical Wounds
Brief Title: Evaluation of the Safety and Efficacy of FBPM10 System in the Treatment of Post-surgical Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KLOX Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-K1002-P011
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Post-surgical Wounds
MeSH Terms: interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with FBPM10 system (Experimental): One breast will be randomized to be treated with FBPM10 System.
  Interventions: Device: FBPM10 System
- Treatment with standard of care (Active Comparator): One breast will be selected to be treated with massages with vitamin E cream.
  Interventions: Other: Massages with vitamin E cream

INTERVENTIONS:
Device: FBPM10 System — Application of the FBPM10 membrane followed by illumination with a multi-Light Emitting Diode (LED) lamp.
  Arms: Treatment with FBPM10 system
Other: Massages with vitamin E cream — The other breast will be treated with wound massages with vitamin E cream.
  Arms: Treatment with standard of care

SUMMARY:
This is a prospective randomized controlled case series in patients having a surgery for bilateral breast reduction. Objectives of the case series are to evaluate the safety and efficacy of the FBPM10 System when compared with standard of care (massages with vitamin E cream) in the treatment of post-surgical wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent form;
2. Female 18 years of age and older;
3. Good general health, stable weight, free of systemic diseases such as diabetes, arthritis, HIV infection or genetic disorder that could influence the outcome of the treatment;
4. Fitzpatrick skin type I to III;
5. Patients with bilateral breast reduction, expected to have newly formed post-surgery breast incisions of comparable length and of comparable appearance, located on comparable skin area;
6. Patients able to understand, willing and able to comply with all study requirements and post-operative instructions.

Exclusion Criteria:

1. Inability to understand the Study and its requirements or to give informed consent;
2. Systemic antibiotic therapy or anti-inflammatory drugs or any other medication(s) that might interfere with healing within the last three months prior to Treatment initiation;
3. Current use of anticoagulants such as (but not limited to) warfarin, clopidogrel, enoxaparin or high doses of aspirin (> 162 mg daily);
4. Female pregnant patient (by medical history or as ascertained by a pregnancy test);
5. Patient with current alcohol use or actively consuming drugs (addiction) as it may interfere with patient's ability to comply with Study procedures;
6. Patient with known photosensitivity, taking drug(s) to treat photosensitivity, with concurrent disease (such as porphyria) or drug(s) (such as methotrexate or chloroquine) known to induce severe photosensitivity of the skin;
7. Patients who are immunocompromised or taking immunosuppressive therapy;
8. Any concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the Study investigational device;
9. Patient has ongoing malignant disease of any type, active systemic, local skin infection or disease, autoimmune disease or any significant chronic disease which, in the opinion of the investigator, might interfere with the evaluation of the Study objectives or would result in non-compliance with the Study protocol;
10. Patients having had surgery in the area to be incised within one year of Study Screening;
11. Patients with tattoos in the areas of incisions;
12. Patients with history or familial history of keloids or hypertrophic scars;
13. Patients with incisions that are actively bleeding;
14. Patients with known skin hypersensitivity;
15. Patients with known allergic reactions to silicone.
16. Patients that cannot start the treatment within 14 days of the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Adverse events, Serious adverse events, device incidents and compliance | Up to 24 weeks
  Number of adverse events, serious adverse events, device incidents and missed treatment visits

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | Up to 24 weeks
  Assessment of the efficacy of FBPM10 and standard of care by the patient and by the investigator via the POSAS
Vancouver Scar Scale (VSS) | Up to 24 weeks
  Assessment of the efficacy of FBPM10 and standard of care by the investigator via the VSS
Ease of wound management | Up to 24 weeks
  Patient's self-assessment of ease of wound management by a specific questionnaire

OTHER OUTCOMES:
External echography | Up to 24 weeks
  Assessment of the aspect and depth of the dermal and epidermal superficial subcutaneous tissues in the two treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Park Medispa, Montreal, Quebec, Canada